CLINICAL TRIAL: NCT03547037
Title: A Phase 1/1b Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of JNJ-63723283, an Anti-PD-1 Monoclonal Antibody, as Monotherapy or in Combination With Erdafitinib in Japanese Subjects With Advanced Solid Cancers
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of JNJ-63723283, an Anti-Programmed Cell Death (PD)-1 Monoclonal Antibody, as Monotherapy or in Combination With Erdafitinib in Japanese Participants With Advanced Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108471; 63723283LUC1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase 1a: JNJ-63723283 (Monotherapy) (Experimental): Participants will receive monotherapy of JNJ-63723283 intravenously. The subsequent dose levels of JNJ-63723283 will be escalated using Bayesian logistic regression model (BLRM).
  Interventions: Drug: JNJ-63723283
- Phase 1b: Erdafitinib Combination (Experimental): Participants will receive erdafitinib in combination with JNJ-63723283 which will be escalated using BLRM.
  Interventions: Drug: JNJ-63723283; Drug: Erdafitinib

INTERVENTIONS:
Drug: JNJ-63723283 — JNJ-63723283 will be administered intravenously.
  Other Names: Cetrelimab
Drug: Erdafitinib — Erdafitinib will be administered orally.
  Arms: Phase 1b: Erdafitinib Combination

SUMMARY:
The primary purpose of this study is to identify the recommended Phase 2 dose (RP2D) of JNJ-63723283 as a monotherapy (Phase 1a part) and to identify the RP2D of JNJ-63723283 when administered in combination with Erdafitinib (Phase 1b part).

ELIGIBILITY:
Inclusion Criteria:

* Radiographically, histologically, or cytologically confirmed advanced or refractory solid tumor(s) that is metastatic or unresectable, and previously received or was ineligible for standard treatment options. Participants with solid tumor(s) for which anti-PD-1 or anti-PD-L1 antibody as a monotherapy is approved in Japan are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Thyroid function laboratory values within normal range
* A woman must be: a) Not of childbearing potential; b) Of childbearing potential and practicing a highly effective, preferably user-independent method of contraception (failure rate of less than (<) 1 percent (%) per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and continue for 5 months following discontinuation of JNJ-63723283 or 3 months following discontinuation of erdafitinib, whichever is longer. Especially participants receiving erdafitinib must agree to use two contraceptive methods and one must be user-independent method; Examples of highly effective contraceptives include: user-independent methods: intrauterine device (IUD) or intrauterine contraceptive system (IUS) and user-dependent methods: combined (estrogen- and progestogen-containing) hormonal contraception or progesterone-containing hormonal contraception. c) Agree not to donate eggs (ova, oocytes), during the study and continue for 5 months following discontinuation of JNJ-63723283 or 3 months following discontinuation of erdafitinib, whichever is longer
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person and must agree not to donate sperm for 5 months following discontinuation of JNJ-63723283 or 5 months following discontinuation of erdafitinib, whichever is longer

Exclusion Criteria:

* Had prior treatment with an anti-PD-1 antibody, anti-PD-L1 antibody or anti-PDL2 antibody within 30 days of first study drug administration and/or has an ongoing Grade 2 or higher immunotherapy-related toxicity. If the subject has an experience of treatment with these agents, the subject must not have had severe immunotherapy-related toxicity
* History of or concurrent interstitial lung disease
* Active autoimmune disease or a documented history of autoimmune disease that requires systemic steroids or immunosuppressive agents
* Grade 3 or higher toxicity effects from previous treatment with immunotherapy
* Has taken immunosuppressive doses of systemic medications, such as corticosteroids doses greater than (>) 10 milligram per day (mg/day) prednisolone or equivalent), within 2 weeks before the planned first dose of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Phase 1a and Phase 1b: Number of Participants with Dose Limiting Toxicity (DLT) | Up to 6 weeks (maximum)
  The DLTs are based on drug-related adverse events and defined as any of the following events: Infusion-related reactions, non-hematologic toxicity of Grade 3 or higher, or certain hematologic toxicity.
Phase 1a and Phase 1b: Severity of DLT as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Up to 6 weeks (maximum)
  Severity of DLT will be graded by using NCI-CTCAE, version 4.03. Severity scale ranges from Grade 1 to Grade 5 with Grades as follows: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), and Grade 5 (Death).

SECONDARY OUTCOMES:
Phase 1b: Number of Participants with Adverse Events and Immune-Related Adverse Event (irAE) by Severity | Approximately up to 3 years
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Severity of Adverse Event will be graded by using NCI-CTCAE, version 4.03. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death) with Grades as follows: Grade 1 (Mild) Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life threatening) and Grade 5 (Death).
Phase 1a and Phase 1b: Number of Participants With Clinically Significant Changes in Vital Signs as a Measure of Safety and Tolerability | Approximately up to 3 years
  Number of participants with clinically significant changes in the vital signs including blood pressure, pulse rate, and body temperature will be reported.
Phase 1a and Phase 1b: Number of Participants With Clinical Laboratory Abnormalities as a Measure of Safety and Tolerability | Approximately up to 3 years
  Number of participants with clinical laboratory abnormalities (clinical laboratory tests include the following: hematology panel, coagulation panel, serum chemistry panel, endocrine panel, serology and pregnancy test [women only]) will be reported.
Phase 1a and Phase 1b: Number of Participants With ECG Abnormalities as a Measure of Safety and Tolerability | Approximately up to 3 years
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Phase 1a and Phase 1b: Maximum Serum Concentration (Cmax) of JNJ-63723283 | Approximately up to 3 years
  The Cmax is the maximum observed serum concentration.
Phase 1a and Phase 1b: Serum Concentration Immediately Prior to the Next Drug Administration (Ctrough) of JNJ-63723283 | Approximately up to 3 years
  Ctrough is the serum concentration immediately prior to the next drug administration of any dose other than the first dose in a multiple dosing regimen.
Phase 1a and Phase 1b: Time to reach Maximum Observed serum Concentration (Tmax) of JNJ-63723283 | Approximately up to 3 years
  The Tmax is defined as actual sampling time to reach maximum observed serum concentration.
Phase 1a and Phase 1b: Area Under the Serum Concentration-Time Curve Between 2 Defined Sampling Points, (t1 and t2) (AUC[t1-t2]) of JNJ-63723283 | Approximately up to 3 years
  The AUC(t1-t2) is the area under the serum concentration-time curve between 2 defined sampling points, t1 and t2.
Phase 1a and Phase 1b: Elimination Half-Life (t1/2) of JNJ-63723283 | Approximately up to 3 years
  T1/2 is the time measured for the serum concentration to decrease by 1 half to its original concentration.
Phase 1a and Phase 1b: Total Systemic Clearance (CL) of JNJ-63723283 | Approximately up to 3 years
  CL is a quantitative measure of the rate at which JNJ-63723283 is removed from the body.
Phase 1a and Phase 1b: Volume of Distribution at Steady-State (Vss) of JNJ-63723283 | Approximately up to 3 years
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution is the apparent volume of distribution at steady-state.
Phase 1b: Cmax of Erdafitinib | Approximately up to 3 years
  The Cmax is the maximum observed plasma concentration.
Phase 1b: Ctrough of Erdafitinib | Approximately up to 3 years
  Ctrough is the plasma concentration immediately prior to the next drug administration of any dose other than the first dose in a multiple dosing regimen.
Phase 1a and Phase 1b: Number of Participants With Anti-JNJ 63723283 Antibodies | Approximately up to 3 years
  Number of participants with anti-JNJ 63723283 antibodies will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa